CLINICAL TRIAL: NCT02774421
Title: Pilot Study of the Effect of Trastuzumab and GM-CSF on Children with Recurrent Ependymoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-1076.cc
Record Dates: First submitted 2016-05-06; First posted 2016-05-17 (Estimated); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Posterior Fossa Ependymoma (PFEPN)
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IT trastuzumab after subQ GM-CSF (Experimental): Patients with localized recurrent PFEPN will be treated with IT trastuzumab following 5-day course of subQ GM-CSF. Surgical resection should be planned (based on institutional surgical scheduling standards) for ideally 2-7 days after IT trastuzumab dosage.
  Interventions: Drug: Trastuzumab after SubQ GM-CSF
- IT trastuzumab in combination with subQ GM-CSF (Experimental): Patients with localized recurrent PFEPN will be treated with IT trastuzumab in combination with GM-CSF to establish a maximum tolerated dosage. GM-CSF will be administered at 250 mcg/m2/dose subQ daily for three (3) days prior to the IT trastuzumab dose.
  Interventions: Drug: Trastuzumab in combination with SubQ GM-CSF

INTERVENTIONS:
Drug: Trastuzumab after SubQ GM-CSF — Administration of trastuzumab following subcutaneous granulocyte-macrophage colony-stimulating factor (GM-CSF). Trastuzumab is a monoclonal antibody targeting HER2-positive cancers, commonly used in breast and gastric cancer treatment.
  Arms: IT trastuzumab after subQ GM-CSF
Drug: Trastuzumab in combination with SubQ GM-CSF — Combine trastuzumab, a monoclonal antibody targeting HER2-positive cancers, with subcutaneous granulocyte-macrophage colony-stimulating factor (GM-CSF). GM-CSF functions as an immune system modulator, promoting the activation and proliferation of dendritic cells, macrophages, and granulocytes.
  Arms: IT trastuzumab in combination with subQ GM-CSF

SUMMARY:
This study plans to detect the presence of trastuzumab by mass spectroscopy in relapsed posterior fossa ependymoma (PFEPN) tumor specimen pre-treated with a single dose of intrathecal (IT) trastuzumab, as well as to evaluate toxicity of intrathecal trastuzumab in combination with subcutaneous (subQ) Granulocyte-macrophage colony-stimulating factor (GM-CSF) in children with relapsed PFEPN

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 months and < 21 years at the time of study enrollment
* Patients must be diagnosed with relapse of previously histologically confirmed PFEPN
* Magnetic resonance (MR) imaging of the brain (performed within 14 days of enrollment) must demonstrate no evidence of diffuse leptomeningeal spread beyond the primary relapse site in posterior fossa and no obstruction of cerebrospinal fluid flow (CSF).
* MR imaging of the total spine (performed within 14 days of enrollment) demonstrates no evidence of spinal metastatic disease.
* Patients must have clinical indication for standard of care surgical resection of relapsed PFEPN tumor for enrollment in Stratum 1
* Patients must meet one of the following performance scores:

  * Eastern Cooperative Oncology Group (ECOG) performance status scores of 0, 1, or 2;
  * Karnofsky score of ≥ 50 for patients > 16 years of age; or
  * Lansky score of ≥ 50 for patients ≤ 16 years of age.
* Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.
* Organ Function Requirements:

  * Adequate Renal Function defined as:

    1) Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥70ml/min/1.73 m2 or 2) A serum creatinine based on age/gender as follows: Maximum Serum Creatinine (mg/dL) Age: Male Female

    1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5

    1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

    ≥ 16 years 1.7 1.4
  * Adequate Liver Function defined as:

    1. Total bilirubin ≤1.5 x upper limit of normal (ULN) for age, and
    2. Serum glutamic oxaloacetic transaminase (SGOT) (AST) or serum glutamate pyruvate transaminase (SGPT) (ALT) < 3 x upper limit of normal (ULN) for age
  * Adequate Bone Marrow Function defined as:

    1. Peripheral absolute neutrophil count (ANC) ≥1,000/µL
    2. Platelet count ≥100,000/µL (transfusion independent)
  * Adequate Cardiac Function defined as:

    1. Shortening fraction > 28% by echocardiogram or
    2. Ejection fraction > 50% by echocardiogram or radionuclide study

Exclusion Criteria:

* Patients with a diagnosis of:

  * spinal cord ependymoma,
  * myxopapillary ependymoma,
  * subependymoma,
  * ependymoblastoma,
  * supratentorial ependymoma, or
  * mixed glioma are NOT eligible for either Stratum.
* Patients with evidence of nodular metastatic spinal disease by MRI are NOT eligible for Stratum 1 but may be eligible for STRATUM 2 if CSF flow is not obstructed based on appropriate imaging studies, and the patient is deemed safe for lumbar puncture by the medical team.
* Patients with clinical contraindications against lumbar puncture are NOT eligible for either Stratum.
* Prior Therapy:

  * Radiation therapy: At least 28 days must have elapsed (at time of starting protocol therapy) since completion of focal radiation therapy for current recurrence for Stratum 2; Patients who have already undergone radiation therapy for current recurrence are NOT eligible for Stratum 1.
  * Myelosuppressive chemotherapy: At least 21 days must have elapsed after the last dose of myelosuppressive chemotherapy; Patients who have been treated with chemotherapy at time of recurrence are NOT eligible for either Stratum.
  * Monoclonal antibodies: At least three (3) half-lives of the antibody must have elapsed since the last dose of a monoclonal antibody (see Appendix I for list of half-lives)
  * Surgical resection: Must have fully healed from any surgical procedure to be safe for lumbar puncture according to treating neurosurgeon and at least 14 days should have elapsed since the surgical procedure.
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are NOT eligible for either Stratum.
* Concomitant Medications

  * Corticosteroids: Patients receiving systemic corticosteroids are NOT eligible for either Stratum.
  * Investigational Drugs: Patients who are currently receiving another investigational drug are NOT eligible for either Stratum.
  * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are NOT eligible for either Stratum.
* Pregnancy, Breast-Feeding, and Contraception

  1. Pregnant or breast-feeding women are NOT eligible. Pregnancy tests must be obtained in females who are post-menarchal.
  2. Women of childbearing potential and male participants with partners of childbearing potential must agree to:

     * use a "highly effective," non-hormonal form of contraception (including abstinence), or
     * two "effective" forms of non-hormonal contraception by the patient and/or partner, and
     * Contraception must continue for the duration of study treatment and for at least seven (7) months after the last dose of study treatment.
* Patients who have an uncontrolled serious infection are NOT eligible for either Stratum.
* Patients who have previously received solid organ transplantation are NOT eligible for either Stratum.
* Patients who have a history of:

  * significant cardiac disease,
  * cardiac disease risk factors, or
  * uncontrolled arrhythmias are NOT eligible for either Stratum.

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Stratum 1: Detection of trastuzumab in tumor following IT administration | 2 weeks
  The presence of trastuzumab will be measured as a binary (yes/no) outcome.
Stratum 2: Determine the Maximum Tolerated Dose (MTD) for IT trastuzumab in combination with fixed doses of subQ GM-CSF | 1 month
  The estimated MTD would be the highest dose at which 0/3 or 1/6 subjects experience a Dose Limiting Toxicity (DLT).

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Macy, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No